CLINICAL TRIAL: NCT02981173
Title: Safety and Efficacy of Psilocybin for the Treatment of Headache Disorders
Brief Title: Psilocybin for the Treatment of Cluster Headache
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: Heffter Research Institute (Other); Ceruvia Lifesciences (Unknown); CH TAC LLC (Unknown)
Responsible Party: Principal Investigator, Deepak C. D'Souza, Professor of Psychiatry, Yale University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 1607018057
Record Dates: First submitted 2016-11-11; First posted 2016-12-05 (Estimated); Last update posted 2023-12-15 (Actual); Status verified 2023-12

CONDITIONS: Cluster Headache
MeSH Terms: conditions — Cluster Headache | interventions — Psilocybin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Psilocybin High Dose (Active Comparator)
  Interventions: Drug: 0.143 mg/kg Psilocybin or 10 mg Psilocybin
- Psilocybin Low Dose (Active Comparator)
  Interventions: Drug: 0.0143 mg/kg Psilocybin or 1 mg Psilocybin
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: 0.143 mg/kg Psilocybin or 10 mg Psilocybin — 0.143 mg/kg psilocybin capsule (weight-based option) or 10 mg psilocybin capsule (fixed-dose option) ingested on each of three test days (5 days apart +/- 1-2 days)
  Arms: Psilocybin High Dose
Drug: 0.0143 mg/kg Psilocybin or 1 mg Psilocybin — 0.0143 mg/kg psilocybin capsule (weight-based option) or 1 mg psilocybin (fixed-dose option) ingested on each of three test days (5 days apart +/- 1-2 days)
  Arms: Psilocybin Low Dose
Drug: Placebo — Microcrystalline cellulose capsule ingested on each of three test days (5 days apart +/- 1-2 days)
  Arms: Placebo

SUMMARY:
The purpose of this study is to investigate the effects of an oral psilocybin pulse regimen in cluster headache. Subjects will be randomized to receive oral placebo, low dose psilocybin, or high dose psilocybin in three experimental sessions, each separated by 5 days. Subjects will maintain a headache diary prior to, during, and after the pulse regimen in order to document headache frequency and intensity before, during, and after the pulse regimen. After at least 6 months from the last experimental session, subjects may be invited for a second round, in which they will be randomized to receive either low dose or high dose psilocybin.

ELIGIBILITY:
Inclusion Criteria:

* Chronic cluster headache with at least one attack daily
* Episodic cluster headache with periods that are predictable and have a duration of approximately 2 months
* Attacks are managed by means involving no more than twice weekly triptan use (e.g., high-flow oxygen, heat/cold pack)

Exclusion Criteria:

* Axis I psychotic disorder (e.g. schizophrenia, bipolar I, depression with psychosis)
* Axis I psychotic disorder in first degree relative
* Unstable medical condition, severe renal, cardiac or hepatic disease, pacemaker, or serious central nervous system pathology
* Pregnant, breastfeeding, lack of adequate birth control
* History of intolerance to psilocybin, lysergic acid diethylamide (LSD), or related compounds
* Drug or alcohol abuse within the past 3 months (excluding tobacco)
* Urine toxicology positive to drugs of abuse
* Use of vasoconstrictive medications (i.e. sumatriptan, pseudoephedrine, midodrine) within five half-lives of test days
* Use of serotonergic antiemetics (i.e. ondansetron) in the past 2 weeks
* Use of antidepressant medications (i.e. amitriptyline, isocarboxazid, fluoxetine, citalopram) in the past 6 weeks
* Use of steroids or certain other immunomodulatory agents (i.e. azathioprine) in the past 2 weeks

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2016-12-05 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-10-21 (Actual)

PRIMARY OUTCOMES:
Time to first attack after completion of pulse regimen | Two months following the completion of pulse regimen (after completion of experimental sessions 1, 2, and 3)
  Measured in days
Time to last attack after completion of pulse regimen | Six months following the completion of pulse regimen (after completion of experimental sessions 1, 2, and 3)
  Measured in days
Change in frequency of attacks | Measured from 2 weeks before to 2 months after completion of pulse regimen using a headache diary
  Average number of attacks (number per week)
Change in intensity of attacks | Measured from 2 weeks before to 2 months after completion of pulse regimen using a headache diary
  Average intensity of attacks (1-10 on visual analog scale)
Change in duration of attacks | Measured from 2 weeks before to 2 months after completion of pulse regimen using a headache diary
  Average duration of attacks (minutes)
Change in cluster period duration compared to typical cluster period (episodic subjects only) | Measured from 2 weeks before pulse regimen to 6 months following the completion of pulse regimen, then comparing to historical average duration of cluster periods
  Duration of cluster period after intervention (days)
Difference in the change in cluster attack frequency between 1st and 2nd round | Measured from 2 weeks before to 2 months after completion for each of the two pulse regimens using a headache diary
  Average number of attacks (number per week); only in those subjects who return for 2nd round
Difference in the change in cluster attack intensity between 1st and 2nd round | Measured from 2 weeks before to 2 months after completion for each of the two pulse regimens using a headache diary
  Average intensity of attacks (1-10 on visual analog scale); only in those subjects who return for 2nd round
Difference in the change in the duration of attacks between 1st and 2nd round | Measured from 2 weeks before to 2 months after completion for each of the two pulse regimens using a headache diary
  Average duration of attacks (minutes); only in those subjects who return for 2nd round

SECONDARY OUTCOMES:
Use of abortive/rescue medication | Measured from 2 weeks before to 2 months after completion of pulse regimen using a headache diary
  Number of times per week
Attack-free time | Measured from 2 weeks before to 2 months after completion of pulse regimen using a headache diary
  Number of 24 hour days (may be nonconsecutive)
Health-Related Quality of life | Measured from 2 weeks before to 2 months after completion of pulse regimen using a headache diary
  Using the CDC's Health-Related Quality of Life (HRQOL) scale
Psychedelic effects | Taken daily on each experimental day after the resolution of psychedelic effects, approximately 6 hours after drug administration
  Using the 5-Dimensional Altered States of Consciousness (5D-ASC) scale
Change in blood pressure | Measured during each experimental session prior to drug administration, every 15 min in the first hour after drug administration, every 30 min in the second hour, and then hourly for 4 hours or until resolution of psychedelic effects (~6 hours post drug)
  Maximum change from baseline during each experimental session (mmHg)
Change in heart rate | Measured during each experimental session prior to drug administration, every 15 min in the first hour after drug administration, every 30 min in the second hour, and then hourly for 4 hours or until resolution of psychedelic effects (~6 hours post drug)
  Maximum change from baseline during each experimental session (beats per minute)
Change in peripheral oxygenation | Measured during each experimental session prior to drug administration, every 15 min in the first hour after drug administration, every 30 min in the second hour, and then hourly for 4 hours or until resolution of psychedelic effects (~6 hours post drug)
  Maximum change from baseline during each experimental session (SpO2)

CONTACTS AND LOCATIONS:
Locations (1):
- VA Connecticut Healthcare System, West Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Schindler EAD, Sewell RA, Gottschalk CH, Flynn LT, Zhu Y, Pittman BP, Cozzi NV, D'Souza DC. Psilocybin pulse regimen reduces cluster headache attack frequency in the blinded extension phase of a randomized controlled trial. J Neurol Sci. 2024 May 15;460:122993. doi: 10.1016/j.jns.2024.122993. Epub 2024 Apr 2. PMID 38581739